CLINICAL TRIAL: NCT00427479
Title: The Prevalence of Oral Allergy Syndrome and Types of Food Commonly Causing Reactions in Birch Pollen Sensitive Patients Who Have Springtime Hayfever
Brief Title: Oral Allergy Syndrome (OAS): a Pilot Study to Evaluate a Clinical Questionnaire as a Diagnostic Tool
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Other Study IDs: 2002UR005B
Record Dates: First submitted 2007-01-26; First posted 2007-01-29 (Estimated); Last update posted 2007-01-29 (Estimated); Status verified 2007-01

CONDITIONS: Rhinitis; Food Allergy
Keywords: Allergy; Food; Hay fever; Screening
MeSH Terms: conditions — Rhinitis; Food Hypersensitivity; Hypersensitivity; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
An increasing number of people have an allergy to birch pollen, which manifests itself as Springtime hayfever. Some will also have cross-reactions to fruits, vegetables and nuts, a condition known as Oral Allergy Syndrome (OAS). Research has demonstrated that the most effective method of diagnosing this problem is by taking a good clinical history and performing skin prick tests using fresh foods.

The aim of the study will be therefore to investigate the prevalence of OAS in a birch-sensitive population using a simple screening tool and establish the range of foods involved. The objective will be to maximise effective treatment for the patients in our large respiratory allergy clinic by using the screening tool to identify patients with OAS and advise them on the usual foods involved. A further objective will be to use the data to discover if there are any patterns of particular foods involved in OAS in UK sufferers.

The study hypotheses are therefore that there is a high prevalence of oral allergy in people with birch pollen allergy; the best way of diagnosing the problem is by using a screening tool and that there is a core set of foods that are commonly involved in OAS in patients seen in the allergy clinic.

DETAILED DESCRIPTION:
Patients will be recruited both prospectively and retrospectively from the Royal Brompton Hospital allergy clinic and through advertisement. Subjects will be identified by diagnosis of birch pollen allergy, either routinely in the RBHT adult allergy clinic or by looking back at patient records. Suitable patients will be invited to participate in the study, with fully informed consent obtained, if they understand written English and fulfil the following criteria:

Criteria for inclusion

* History of Springtime hayfever
* Positive skin prick test (  3mm) to Birch
* FEV1.> than 70% predicted or greater than 1.5L
* Aged 16 years or more

Exclusion criteria

* Pregnancy
* Existing medical condition which could be affected by a severe response on challenge
* Aged under 16
* FEV1.< than 70% predicted or greater than 1.5L

On recruitment

After a full explanation of the study given, patients who agree to participate will be asked to sign the consent form, a copy of which will be placed in the medical notes, and a second copy sent to the Ethics Committee Administrator. Participants will then be booked in for visit one and advised to avoid short acting antihistamines for 72 hours and long acting ones for a week, prior to their prick prick test.

The OAS screening tool will be completed for every patient. A venous blood sample will be taken and stored for the measurement of total IgE and specific IgE RAST tests for birch, apple, celery and hazelnuts. A questionnaire will be completed by the patient assessing the effect any food reactions is having on their diet and social life. The researcher will then complete a 24-hour food recall questionnaire with the patient, to ascertain their normal dietary intake.

The patient will then be asked whether they have taken anti-histamines in the last 72 hours, and if they have not then prick prick tests can be performed using a range of different fresh fruits, vegetables, nuts and Birch and Grass reagent. The tests will be undertaken according to EAACI recommendations, with a positive and negative control. The allergen content of fresh foods is unknown, but using data from previous studies, a wheal of 3mm will be considered positive, and a wheal of 5 mm strongly positive.

All participants will then be invited to return to undergo one single blind, placebo food challenge. Those classed as negative responders will then undergo two double blind, placebo-controlled food challenges (DBPCFC), one being an active substance and one a control substance. Following these challenges, those still classed as negative responders will undergo an open challenge with the active substance. The only exclusion criteria will be those subjects who have previously reported an anaphylactic response to the active challenge material.

ELIGIBILITY:
Inclusion Criteria:

* History of Springtime hayfever
* Positive skin prick test (  3mm) to Birch
* FEV1 > than 70% predicted or greater than 1.5L
* Aged 16 years or more

Exclusion Criteria:

* Pregnancy
* Existing medical condition which could be affected by a severe response on challenge
* Aged under 16
* FEV1 < than 70% predicted or greater than 1.5L

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2002-07; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Isabel J Skypala, BSc, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton & Harefield NHS TRust, London, United Kingdom